CLINICAL TRIAL: NCT03605173
Title: Free Vitamin D Correlate Better With BMD and Fracture Than Total Serum Vitamin D?
Brief Title: Study on the Correlation of Free Vitamin d With BMD and Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Limin Rong (Other)
Responsible Party: Sponsor-Investigator, Limin Rong, professor, department of spine surgery, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: free vitamin d - bmd
Record Dates: First submitted 2018-07-01; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- free vitamin d (Experimental): free vitamin is directly measured from blood serum using an ELISA kit
  Interventions: Diagnostic Test: free vitamin d test
- total vitamin d (Experimental): Total vitamin d is measured routinely from blood serum
  Interventions: Diagnostic Test: total vitamin d

INTERVENTIONS:
Diagnostic Test: free vitamin d test — using the patient's blood serum ELISA test for free vitamin d can be performed
  Arms: free vitamin d
Diagnostic Test: total vitamin d — routinely measured from serum
  Arms: total vitamin d

SUMMARY:
According to the free hormone hypothesis, the biological activity of a hormone is carried by the portion that is not bound to protein or its carrier in circulation. Based on this, we believe that the free vitamin d, which is the proportion of Vitamin D unbound to vitamin D binding protein and albumin, performs the calcium-regulating functions of the vitamin. Hence, our objective is to study whether free vitamin correlated better with BMD and fracture than the total vitamin D.

DETAILED DESCRIPTION:
Osteoporosis is a major health issue worldwide as it increases the risk of fragility fracture and chronic disability. The studies on the association between vitamin d and osteoporosis have yielded conflicting results. While some have shown a positive correlation, others have concluded that there is no association at all. Recent reports have shown vitamin D supplementation do not prevent fragile fractures. This might be because the actual vitamin D status, which should be the free vitamin D, has not been measured.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of osteoporosis and with or without fracture
* post- menopausal women
* age > 48 years

Exclusion Criteria:

* vitamin D supplementation in recent 6 months
* patients on steroid
* age < 48 years
* patients with chronic diseases such as liver cirrhosis, renal failure, hypertension, hyperparathyroidism

Min Age: 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Free vitamin D | ! day
  measured using free vitamin D Elisa kit
Total vitamin D | ! day
  It is measured as a part of routine investigation at the time of admission

SECONDARY OUTCOMES:
BMD | ! day
  Bone mineral density is measured using the Dual-energy X-ray absorptiometry
Vertebral fracture | ! day
  With the help of plain X-ray

CONTACTS AND LOCATIONS:
Overall Officials: Kishor Chhantyal, MBBS, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third affiliated hospital of sun yat sen university, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chhantyal K, He L, Mo J, Yin M, He T, Chen Y, Yang Y, Zhang L, Rong L. Free vitamin D correlate better with bone mineral density and thoracolumbar junction osteoporotic vertebral fractures than serum vitamin D. BMC Musculoskelet Disord. 2020 Mar 12;21(1):164. doi: 10.1186/s12891-020-3179-7. PMID 32164704